CLINICAL TRIAL: NCT01229397
Title: A Phase III Open, Randomized, Parallel, Multi-center Study in Children Aged 6 - 35 Months to Compare the Immunogenicity and Safety of a Single 0.5 mL Dose of Inflexal V With a 0.25 mL 2-dose Regimen of Inflexal V Administered According to a 0/4 Week Schedule
Brief Title: Immunogenicity and Safety of a Single 0.5 mL Dose of Inflexal V With a 0.25 mL 2-dose Regimen of Inflexal V
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INF-V-A005
Record Dates: First submitted 2010-10-22; First posted 2010-10-27 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Immunisation
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Inflexal V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inflexal V 0.25 mL x 2 (Active Comparator)
  Interventions: Biological: Inflexal V
- Inflexal V 0.5 mL x 1 (Experimental)
  Interventions: Biological: Inflexal V

INTERVENTIONS:
Biological: Inflexal V — vaccination with Inflexal V 0.25 mL administered twice, 4 weeks apart
  Arms: Inflexal V 0.25 mL x 2
Biological: Inflexal V — Inflexal V 0.5 mL administrated once only
  Arms: Inflexal V 0.5 mL x 1

SUMMARY:
The study aims to evaluate the immunogenicity of a single full (0.5 mL) dose and a 0.25 mL 2-dose regime of Inflexal V in unprimed children aged 6 - <36 months, using the EMA guideline for the re-registration of the seasonal influenza vaccine in adults (aged ≥18 ≤60 years) as reference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children
* Aged ≥6 to <36 months on Day 1
* Born at a gestational age ≥37 weeks
* Written informed consent
* No previous influenza vaccination

Exclusion Criteria:

* Acute respiratory infection or other acute disease
* Acute febrile illness (≥38.0 °C)
* Past vaccination with an influenza vaccine, including vaccination against the influenza strain A/California/7/2009 (H1N1)-like virus
* Laboratory-confirmed infection with any influenza strain, including the pandemic influenza strain H1N1 (A/California/7/2009 (H1N1)-like virus)
* Known hypersensitivity to any vaccine component
* Known history of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, incl. oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent for ≥14 days (inhaled or topical steroids are allowed)
* Known immunodeficiency (including leukemia, cancer, HIV seropositivity)
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Vaccination with the MMR vaccine in the past 4 weeks, or planned within the study period
* Participation in another clinical trial
* Child or legal charge of the investigator or an employee at the study site, or living in the same household as the investigator/employee and/or dependent on the investigator/employee
* Suspected non-compliance

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Principi, Prof Dr, Principal Investigator — Institute of Paediatrics, University of Milan, Fondazione IRCCS "Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena", Via Commenda 9, 20122, Milano, Italy; Gian Vincenzo Zuccotti, Prof Dr, Principal Investigator — Department of Pediatrics, Department of Clinical Sciences, Università di Milano, L. Sacco Hospital, 74, Via GB Grassi,
Locations (2):
- Italy (2):
  - Department of Pediatrics, Department of Clinical Sciences, Università di Milano, L. Sacco Hospital, Milan
  - Institute of Paediatrics, University of Milan, Fondazione IRCCS "Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena", Milan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 05 October - 17 January 2011; Location: University of Milan
Groups:
- Inflexal V 0.25 mL x 2: 2 doses of Inflexal V influenza vaccine (surface antigen, inactivated, virosome) 2010/2011, 4 weeks apart, containing per 0.25 mL dose:
  * 7.5 μg HA antigen of A/California/7/2009 (H1N1)-like virus
  * 7.5 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus
  * 7.5 μg HA antigen of B/Brisbane/60/2008-like virus
- Inflexal V 0.5 mL x 1: 1 dose of Inflexal V influenza vaccine (surface antigen, inactivated, virosome) 2010/2011, containing per 0.5 mL dose:
  * 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus
  * 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus
  * 15 μg HA antigen of B/Brisbane/60/2008-like virus
Period: Overall Study
Arm/Group | Inflexal V 0.25 mL x 2 | Inflexal V 0.5 mL x 1
Started | 103 | 102
Completed | 92 | 93
Not Completed | 11 | 9
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 7 | 6
Not completed — Migrated/moved from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inflexal V 0.25 mL x 2: Two 0.25 mL doses (on Day 1 and 29)
- Inflexal V 0.5 mL x 1: One 0.5 mL dose (on Day 1)
- Total: Total of all reporting groups
Arm/Group | Inflexal V 0.25 mL x 2 | Inflexal V 0.5 mL x 1 | Total
Number analyzed (Participants) | 103 | 102 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 103 | 102 | 205
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.8 (0.52) | 1.8 (0.61) | 1.8 (0.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 66 | 65 | 131
Region of Enrollment [Number; unit: participants]
  Italy | 103 | 102 | 205

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of a Single Full (0.5 mL) Dose and a 0.25 mL 2-dose Regimen of Inflexal V, Using the EMA Guideline for the Re-registration of the Seasonal Influenza Vaccine in Adults (Aged ≥18 to ≤60 Years) as Reference
Description: Seroprotection rate
Time Frame: This assesment was done for immunogenicity data collected at Day 29 after completion of designated vaccination regimen
Population: Intention to treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage subjects
Arm/Group | Inflexal V 0.25 mL x 2 | Inflexal V 0.5 mL x 1
Number analyzed (Participants) | 98 | 99
percentage subjects
  Percentage of subjects seroprotected: A/H1N1 | 99.0 [94.4 to 100] | 98.0 [92.9 to 99.8]
  Percentage of subjects seroprotected: A/H3N2 | 99.0 [94.4 to 100] | 97.0 [91.4 to 99.4]
  Percentage of subjects seroprotected: B-strain | 92.2 [85.8 to 97.1] | 86.9 [78.6 to 92.8]

2. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events as a Measure of Safety and Tolerability
Time Frame: Solicited local and systemic AEs were collected from Day 1 (day of vaccination) to Day 4 inclusive using a subject diary
Population: Safety population, all vaccinated subjects
Measure: Number; unit: participants
Arm/Group | Inflexal V 0.25 mL x 2 - After 1st Vaccination | Inflexal V 0.25 mL x 2 - After 2nd Vaccination | Inflexal V 0.5 mL x 1
Number analyzed (Participants) | 102 | 101 | 100
participants
  AEs (unsolicited and solicited) | 51 | 48 | 49
  Unsolicited AEs | 29 | 32 | 30
  Solicited local AEs | 22 | 16 | 17
  Solicited systemic AEs | 16 | 16 | 20

3. Primary Outcome: Immunogenicity of a Single Full (0.5 mL) Dose and a 0.25 mL 2-dose Regimen of Inflexal V, Using the EMA Guideline for the Re-registration of the Seasonal Influenza Vaccine in Adults (Aged ≥18 to ≤60 Years) as Reference
Description: Seroconversion rate
Time Frame: This assesment was done for immunogenicity data collected at Day 29 after completion of designated vaccination regimen
Population: Intention to treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage subjects
Arm/Group | Inflexal V 0.25 mL x 2 | Inflexal V 0.5 mL x 1
Number analyzed (Participants) | 98 | 99
percentage subjects
  Percentage of subjects seroconverted: A/H1N1 | 92.9 [85.1 to 97.3] | 95.5 [88.8 to 98.7]
  Percentage of subjects seroconverted: A/H3N2 | 99.0 [94.4 to 100] | 97.0 [91.4 to 99.4]
  Percentage of subjects seroconverted: B-strain | 92.9 [85.8 to 97.1] | 86.9 [78.6 to 92.8]

4. Primary Outcome: Immunogenicity of a Single Full (0.5 mL) Dose and a 0.25 mL 2-dose Regimen of Inflexal V, Using the EMA Guideline for the Re-registration of the Seasonal Influenza Vaccine in Adults (Aged ≥18 to ≤60 Years) as Reference
Description: GMT-fold increase - calculated as the GMT on Day 22 divided by the baseline GMT value
Time Frame: This assesment was done for immunogenicity data collected at Day 29 after completion of designated vaccination regimen
Population: Intention to treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: Fold (ratio)
Arm/Group | Inflexal V 0.25 mL x 2 | Inflexal V 0.5 mL x 1
Number analyzed (Participants) | 98 | 99
Fold (ratio)
  GMT fold increase from baseline: A/H1N1 | 25.5 [21.3 to 30.5] | 19.6 [16.9 to 22.7]
  GMT fold increase from baseline: A/H3N2 | 31.6 [26.7 to 37.3] | 24.6 [20.7 to 29.3]
  GMT fold increase from baseline: B-strain | 12.8 [11.2 to 14.6] | 14.7 [12.3 to 17.4]

ADVERSE EVENTS:
Time Frame: Any AE occurring within 1 month (minimum 28 days) following vaccine administration was recorded. Any SAE occurring from study start up to 6 months (at least 180 days) following vaccine administration was recorded.
Arm/Group | Inflexal V 0.25 mL x 2 - After 1st Vaccination | Inflexal V 0.25 mL x 2 - After 2nd Vaccination | Inflexal V 0.5 mL x 1
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/101 | 5/100
Other Adverse Events (participants affected / at risk) | 51/102 | 48/101 | 49/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inflexal V 0.25 mL x 2 - After 1st Vaccination (N=102) | Inflexal V 0.25 mL x 2 - After 2nd Vaccination (N=101) | Inflexal V 0.5 mL x 1 (N=100)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenterisits rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inflexal V 0.25 mL x 2 - After 1st Vaccination (N=102) | Inflexal V 0.25 mL x 2 - After 2nd Vaccination (N=101) | Inflexal V 0.5 mL x 1 (N=100)
Pyrexia (General disorders) | 8 (8) | 11 (11) | 15 (15)
Pyrexia (General disorders) | 11 (11) | 10 (13) | 9 (9)
Erythema (at the injection site) (General disorders) | 15 (15) | 7 (7) | 10 (10)
Induration (at the injection site) (General disorders) | 7 (7) | 2 (2) | 6 (6)
Pain (at the injection site) (General disorders) | 11 (11) | 10 (10) | 9 (9)
Haemorrhage (at the injection site) (General disorders) | 3 (3) | 4 (4) | 5 (5)
Malaise (General disorders) | 9 (9) | 8 (8) | 7 (7)
Otitis media acute (Infections and infestations) | 4 (4) | 3 (3) | 5 (5)
Rhinitis (Infections and infestations) | 1 (1) | 9 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 60 days from the time submitted to the sponsor for review. The sponsor reserves the right to remove any proprietary or confidential information and to require that publication be delayed for up to 60 additional days to enable the sponsor to prepare and file patent applications.